CLINICAL TRIAL: NCT06375538
Title: Ultrasound Evaluations of Diaphragm and Intercostal Muscle to Predict the Failure of High-Flow Nasal Cannula Therapy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2022-527
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: High-flow Nasal Cannula; Ultrasound Evaluation; Diaphragm and Intercostal Muscle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to predict the failure of High-flow Nasal Cannula oxygenation therapy by ultrasound evaluation of diaphragm and intercostal muscle contraction during the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* needing High-flow Nasal Cannula oxygenation therapy

Exclusion Criteria:

* received mechanical ventilation, including invasive or noninvasive ventilation within one month prior to enrollment
* history of neuromuscular disorders (e.g., myasthenia gravis, Guillain-Barre syndrome);
* immediate endotracheal intubation is required (life-threatening hypoxemia)
* extensive damage to the thoracic skin (e.g., burns) unable to undergo ultrasonography
* pregnancy
* attending physician deemed it inappropriate to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 who are admitted to ICU will be screened for eligibility.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound evaluation of diaphragm | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  Thickness of the diaphragmatic muscle and the diaphragm thickening fraction (DTF) by ultrasound evaluation
Ultrasound evaluation of intercostal muscle movement index | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  the parasternal intercostal muscles thickening fraction by ultrasound evaluation
The patient's condition deteriorated and required noninvasive or intubated invasive mechanical ventilation. | up to 30 days after High-flow Nasal Cannula (HFNC)oxygenation therapy.
  Failing or not failing HFNC, the rate of needing noninvasive or intubated invasive mechanical ventilation.

SECONDARY OUTCOMES:
ICU stay | up to one month after High-flow Nasal Cannula (HFNC)oxygenation therapy.
  patients enrolled will be followed for length of ICU stay
Hospital stay | up to one month after High-flow Nasal Cannula (HFNC)oxygenation therapy.
  patients enrolled will be followed for length of Hospital stay
all cause mortality | up to one month after High-flow Nasal Cannula (HFNC)oxygenation therapy.
  all cause mortality
Oxygen saturation | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  Oxygen saturation
respiratory rate | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  respiratory rate
oxygen concentration | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  oxygen concentration
flow velocity of HFNC | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  flow velocity of HFNC
VT | Six times a day by the 0,2,6,12,18,24 hours following initiation of High-flow Nasal Cannula (HFNC)oxygenation treatment.
  VT
duration on HFNC | up to one month
  patients enrolled for the duration of HFNC

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China